CLINICAL TRIAL: NCT06345807
Title: Innovative Care Pathway in Physical Activity and Behavior Change in Coronary Patients Post Cardiac Rehabilitation
Brief Title: Innovative Care Pathway in Physical Activity and Behavior Change in Coronary Patients Post-cardiac Rehabilitation
Acronym: APIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-A02617-38
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Individualised Physical Activity Program; Coronary Patient
Keywords: cardiac rehabilitation; ischemic heart disease; physical activity; wearables
MeSH Terms: conditions — Myocardial Ischemia; Motor Activity | interventions — Commission on Professional and Hospital Activities

STUDY DESIGN:
Intervention Model Description: interventional study, randomized in 3 parallel groups, single center,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized physical activity program (Experimental)
  Interventions: Other: Individuals activity programs
- Physical Activity program defined without optimisation (Active Comparator)
  Interventions: Other: activity program
- no Physical Activity program (Other)
  Interventions: Other: no Physical Activity program

INTERVENTIONS:
Other: Individuals activity programs — activity program will be adjusted every week by practitioner for each patient following data coming from the wearable device ( connected whatch and bellt for 12 months)
  Arms: Individualized physical activity program
Other: activity program — pre established program without adjustement. The patient has connected whatch and bellt for 12 months
  Arms: Physical Activity program defined without optimisation
Other: no Physical Activity program — no Physical Activity (PA)program but just PA recommendations.PA is carried out independently (common practice).The patient has connected whatch and bellt for 12 months
  Arms: no Physical Activity program

SUMMARY:
The objective of this 18-month research is to show the effectiveness of an individualized physical activity( PA) compared to standard PA management and voluntary PA, to achieve a change in the behavior of the coronary patient.

ELIGIBILITY:
Inclusion Criteria:

* Post-infarction coronary artery patient aged 18 years and older, with no gender difference.
* Patients engaged in a follow-up care and cardiovascular rehabilitation program at the Supervaltech center.
* Patient at low to moderate RARE risk of complication (RARE score 2 to 3)
* Patients equipped with smartphones, laptops or other equipment compatible with downloading an application with their personal ID
* Patient able to understand French for the purpose of conducting the study.
* Affiliated member or beneficiary of a social security scheme.
* Participant who has been informed and has given free, informed and written consent (no later than the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Patients with a formal contraindication to physical activity such as: unstabilized coronary syndrome, decompensated heart failure, severe ventricular arrhythmias, intracardiac thrombus at risk embolic, PAH, moderate pericardial effusion, history of thrombophlebitis with or without pulmonary embolism, severe and/or symptomatic left ventricular ejection obstruction.
* Patients with ongoing infectious disease
* Participant whose physical and/or psychological health is severely impaired, which in the opinion of the investigator may affect the study participant's compliance.
* Participant included in other research
* Participant in a period of exclusion from another research still in progress at the time of inclusion.
* Protected participant: an adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.
* Pregnant, breastfeeding or parturient women.
* Participant hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
6 minutes walk test | 18 months
  patient behaviour change measured with the six minute walk test distance

CONTACTS AND LOCATIONS:
Overall Officials: Deva BAS, MD, Principal Investigator — Clinique SSR SuperValtech

IPD SHARING:
Plan to Share IPD: No